CLINICAL TRIAL: NCT05774964
Title: A Prospective, Single-arm, Single-center, Phase II Clinical Trial to Evaluate the Efficacy of Quintuple Method for the Treatment of Multiple Refractory Colorectal Liver Metastases
Brief Title: Quintuple Method for Treatment of Multiple Refractory Colorectal Liver Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230303zzg
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: For Patients With Colorectal Cancer Liver Metastases Who Were Not Able to Curative Surgical Resection.Focused on the Treatment Effect With the Quintuple Method
Keywords: Quintuple method; Colorectal Liver Metastases
MeSH Terms: interventions — Oxaliplatin; S 1 (combination); Tegafur; gimeracil; Cetuximab; Metronidazole; Vitamin A; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chemotherapy alone group (Experimental): Patients treated with chemotherapy using SOX regimen alone. SOX regimen every 3 weeks,oxaliplatin via intravenous drip on d1 at a dose of 130 mg/m2 × patient 's body surface area, and tegafur orally on d2-d15 at 20 mg three times daily.
  Interventions: Drug: Oxaliplatin; Drug: S1
- Chemotherapy targeted group (Experimental): Patients treated with cetuximab targeted therapy in combination with chemotherapy using SOX regimen.SOX regimen every 3 weeks, oxaliplatin via intravenous drip on d1 at a dose of 130 mg/m2 × patient 's body surface area, and tegafur orally on d2-d15 at 20 mg three times daily. Cetuximab combined with chemotherapy was administered simultaneously,once every three weeks, and intravenous drip was performed before oxaliplatin at a dose of 250 mg/m2 × body surface area.
  Interventions: Drug: Oxaliplatin; Drug: S1; Drug: Cetuximab
- Quintuple method group (Experimental): Patients treated with a combination of SOX regimen, cetuximab, and folic acid, vitamin A, and metronidazole three-drug regimen.SOX regimen every 3 weeks, oxaliplatin via intravenous drip on d1 at a dose of 130 mg/m2 × patient 's body surface area, and tegafur orally on d2-d15 at 20 mg three times daily. Cetuximab combined with chemotherapy was administered simultaneously,once every three weeks, and intravenous drip was performed before oxaliplatin at a dose of 250 mg/m2 × body surface area. Metronidazole 0.4g/time, qd;vitamin A 5,000 units/time, qd; folic acid 5 mg/time,qd. The latter three drugs were continued until the end of all chemotherapy cycles.
  Interventions: Drug: Oxaliplatin; Drug: S1; Drug: Cetuximab; Drug: Metronidazole; Drug: Vitamin A; Drug: Folic acid

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin via intravenous drip on d1 at a dose of 130 mg/m2 × patient 's body surface area
Drug: S1 — Orally on d2-d15 at 20 mg three times daily
  Other Names: Tegafur,Gimeracil and Oteracil Porassium Capsules
Drug: Cetuximab — Cetuximab combined with chemotherapy was administered simultaneously, once every three weeks,and intravenous drip was performed before oxaliplatin at a dose of 250 mg/m2 × body surface area.
  Arms: Chemotherapy targeted group; Quintuple method group
Drug: Metronidazole — Metronidazole 0.4g/time, qd
  Arms: Quintuple method group
Drug: Vitamin A — Vitamin A 5,000 units/time, qd
  Arms: Quintuple method group
Drug: Folic acid — Folic acid 5 mg/time, qd
  Arms: Quintuple method group

SUMMARY:
The aim of this study is to explore the therapeutic effect of Quintuple method in the treatment of patients with multiple and refractory liver metastases from colorectal cancer. A randomized single-arm clinical trial was conducted.The intervention group was treated with single SOX chemotherapy, SOX chemotherapy combined with cetuximab targeted therapy, SOX chemotherapy combined with low-dose cetuximab targeted therapy combined with three-drug regimen（Quintuple method）, and the RECIST 1.1 solid tumor evaluation criteria were used to assess the disease.

DETAILED DESCRIPTION:
Patients with inoperable colorectal liver metastases were selected for genetic testing and enrolled if Kras/Nras/Braf wild-type was detected. The enrolled patients were randomly divided into three groups, in which patients in the single chemotherapy group were treated with SOX regimen alone for chemotherapy;patients in the chemotherapy targeted group were treated with SOX regimen chemotherapy combined with cetuximab targeted therapy; patients in the Quintuple method group were treated with SOX regimen chemotherapy,cetuximab targeted therapy and folic acid, vitamin A, and metronidazole three-drug regimen. Specific drugs were administered at the following doses: SOX regimen every 3 weeks, oxaliplatin via intravenous drip on d1 at a dose of 130 mg/m2 × patient 's body surface area, and S1 orally on d2-d15 at 20 mg three times daily. Cetuximab combined with chemotherapy was administered simultaneously, once every three weeks, and intravenous drip was performed before oxaliplatin at a dose of 250 mg/m2 × body surface area. Metronidazole 0.4 g/time, qd; vitamin A 5,000 units/time, qd; folic acid 5 mg/time, qd. The latter three drugs were continued until the end of all chemotherapy cycles.Tumor markers associated with liver metastases from colorectal cancer,including magnetic resonance imaging and computed tomography, wererepeated every 3 months and disease was assessed using RECIST 1.1 criteria for the evaluation of solid tumors. The primary end point was death, and the secondary end point was disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years at the time of signing the informed consent form;
2. Patients with histologically or cytologically confirmed adenocarcinoma of the colon or rectum (stage IV);
3. Patients with liver metastases found by imaging examination, and liver metastases cannot be radically resected, Or relapse liver metastasis;
4. At least one measurable metastatic lesion as defined by RECIST version 1.1;
5. Genetic test results are Kras/Nras/Braf wild-type or mutation type;
6. ECOG performance status 0-1;
7. Except for the liver, other organs function well;
8. Willingness and ability to comply with scheduled visits, treatment plans,laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients with non-primary intestinal cancer;
2. Patients whose primary tumor as well as metastases can be radically resected by surgery;
3. One or several serious allergies to each drug required for the trial;
4. Combined with respiratory, circulatory, urinary, hematopoietic and other serious underlying diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 2 years
  Overall response rate (ORR) is defined as the proportion of patients with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1
Overall Survival (OS) | Up to approximately 2 years
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up. For subjects who survived or were lost to follow-up by the data analysis cutoff date, survival was truncated by the subject's last known survival time
Progression Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of randomization to the date of the first documented progression or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Liaoning Tumor Hospital & Institute, Shenyang, Liaoning, China